CLINICAL TRIAL: NCT03185689
Title: Effect of Diabetic Self-management Education (DSME) on Clinical, Psychosocial, and Behavioral Outcomes Among People With Type 2 Diabetes Attending Jimma University Medical Center (JUMC)
Brief Title: Diabetes Self-Management Education (DSME) and Its Effect on Clinical, Psychosocial, and Behavioral Outcomes
Acronym: DSME-Et
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Fikadu Balcha Hailu, Principal Investigator, Jimma University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DSME-Et
Record Dates: First submitted 2017-05-27; First posted 2017-06-14 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycemic control; Diabetes self-management education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: DSME is model assumed to empower diabetes patients in the area of self-care practice. To bring this behavioral change it has been hypothesized that an intensified DSME which is given in organized, interlinked and supported by take home activities is effective in glycemic control. As a teaching material, illustrative booklet was prepared in two local languages. Similarly, fliers have been given following each DSME session. Specifically for educational sessions, copy of the booklet was prepared in larger posters. The education is not only one way type of education, rather there have been a vast experience sharing among the patient, whether they have been doing in the recommended way or not. Then the facilitator educate them what is right and recommended. Local culture, values and beliefs were taken into account on each of the sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Effectiveness of an intensified DSME in T2D adult patients
  Interventions: Behavioral: Effectiveness of an intensified DSME in T2D adult patients
- Comparison group (No Intervention): The comparison group have got the usual traditional way of education, which is given occasionally for all of diabetes patients at waiting area. Other than this, the comparison group didn't get an organized and intensified DSME.

INTERVENTIONS:
Behavioral: Effectiveness of an intensified DSME in T2D adult patients
  Arms: Intervention group

SUMMARY:
In relation to rapid urbanization, demographic transition and childhood conditions obesity and type 2 diabetes (T2D) is increasing in an alarming rate in Africa. With an increase in the rate of diabetes in Ethiopia, responses to reduce its occurrence and delaying or preventing complications is not adequate. One of these strategies is empowerment of diabetes patients on self-care.

The main objective of this project is to assess effects of phased and intensified DSME on psycho-social, clinical, and behavioral outcomes among adults with T2D in Ethiopia.

An interventional two groups study design was employed to determine the desired effect of DSME. The study participants were selected randomly from adult T2D patients attending Jimma University Medical Center (JUMC) chronic illness follow-up clinic. Using the assumption of increasing the proportion of people with controlled blood glucose from 18% to 33% the sample was calculated 120 with participants in the intervention group and 120 in the comparison group.

To reduce risk of contamination, we planned to vary the intervention and the comparison group based on their residence using kebele (the smallest administrative unit) for residents of Jimma town and woreda or district for those outside of Jimma town. Because of the inconvenience to vary days of appointment, where those supposed to come on Monday were coming on Tuesday and those supposed to come on Monday were coming on Tuesday, that created a high risk of mix-up of participants. Because of this reason, though the baseline was collected from February 2016 to May 2016, the intervention was delayed by five months and then started on November.

Face to face group-based DSME has been given to the intervention group from November 2016 to April 2017. Then the participants will be further followed for three months to determine the effect of phased and intensified DSME on the control of BGL as measured by HbA1c.

In order to make it culture-friendly educational materials were prepared with two widely used languages, Amharic and Afan Oromoo. First, the teaching materials were prepared in English then translated to Amharic and Afan Oromoo separately by bilingual experts. Then, different bilingual experts back translated to English. Finally, with these experts, common discussion was made and the final teaching materials were produced. The package of teaching materials includes booklets, fliers, and posters prepared in both languages.

DETAILED DESCRIPTION:
As incidence and prevalence of non-communicable chronic diseases (NCDs) is increasing, care of individuals with NCDs become challenging, complex and expensive (1). One of the models used for the management of NCDs is the mode developed by Wagner and his colleagues in 1990s. Of the six components of the model self-management support has been identified and customized to diabetic care which helps to assist diabetic patients to overcome attitudinal and motivational barriers, improve their self-management skills and feelings of self-efficacy (2).

The objective of DSME is to support the individual to make informed decision, cope with daily demands of diabetes, make behavioral changes that support their self-care practice, active collaboration with the health care team and improve clinical outcomes, health status, and quality of life (3, 4).

In some of developed countries, it was found that DSME is effective in reducing HbA1c, BGL, BP, BMI, anxiety, need for diabetes medication and risk of complications as well as improve diabetes knowledge, sound activity, diet, self-care practice, quality of life (5-8).

Though very few intervention studies related to DSME are conducted in a very few countries (9-12), the role of culture friendly DSME in Africa is not well understood. In addition, since Africa has a different living style, culture, belief, and probably different risk factors of diabetes as well, the effectiveness of DSME is not well understood and it has not been given a due attention. Similarly, in Ethiopia despite large number of people with diabetes, so far to our knowledge no organized DSME has been developed, tested and implemented.

Therefore, exploring effectiveness of DSME in Ethiopian context is paramount. The findings from this study can be important to help patients living with Diabetes 2 to leave healthier life by reducing/preventing the occurrence of complications. Moreover, it may initiate policy makers, health planners and other relevant stakeholders about importance of diabetes control using self-management education and support. At the same time, self-management is expected to contribute to improve clinical outcome, reduce risk factors, prevent or delay of disabilities and ultimately improve the quality of life for the individuals and their families. This may in turn enables societal members to participate in the country's economic growth and development. The findings of this study will also be used as a baseline for future related studies. The finding of the study can also be used as a starting point for the Ethiopian Federal Ministry of Health (FMoH) and the respective regional health bureaus to develop and implement culturally friendly DSME model. Moreover, it can initiate relevant bodies to design short-term and long-term curriculum for training of relevant front line health care providers, like nurses or community health workers, who will have a central role in the support of clients with diabetes.

Objective The main objective of the project is to assess effects of DSME on behavioral (self-care practice including nutrition and activity, medication adherence and healthcare utilization), clinical (glycemic control as measured by HbA1c, BP, BMI, and WC) and psychosocial (HRQoL, depression, anxiety, self-efficacy and diabetes knowledge,) outcomes among adults with T2D in Ethiopia, and particularly in Jimma zone.

Research questions

1. How do DSME affect dietary choices and exercise among adults with T2D attending JUMC chronic illness follow-up clinic?
2. Do DMSE improve medication adherence and health care utilization by adults with T2D attending JUMC chronic illness follow-up clinic?
3. Do DSME improve the health status of adults with T2D attending JUMC chronic illness follow-up clinic? These research questions will be addressed in separate sub studies. Taking glycemic control as primary outcome, the effectiveness of DSME will be evaluated by an absolute increase of the proportion of people with good glycemic control by 15%.

Design A before and after interventional controlled study design will be employed to explore the effects of DSME among adults with T2D attending JUMC.

Setting The study will be conducted in JUMC, Jimma Ethiopia. Currently 477 T2D patients get follow-up care in the chronic diseases follow up clinic of the hospital. Of these around 330 of them are 18 years and above. So far, to our knowledge there is no formal structured education arrangement for all diabetes patients visiting the clinic.

Study period The project will be completed within four years period from January 2015 through 2018.

Recruitment, participants and sampling Based on physicians' diagnoses recorded and history of medicines they are taking T2D patients were identified. Further, these T2D patients were categorized according to their living residence. Roughly, since the number of patients from kebeles (the smallest administrative unit) of Jimma town and woredas/districts outside of Jimma town is equal, kebele for those from Jimma town and woreda for those from outside of Jimma town were used for patient categorization. Then based on their kebele/woreda block randomization to either the intervention or the comparison group was made. For monitoring participation in the DSME sessions, on recruitment their full address was collected.

Sample size was calculated using Epi info_7.exe. with the assumption that DSME will increase the proportion of diabetic patients with controlled BGL from 18% (13) to 33%. Adding 15% non-response rate the final sample size become 240, where 120 are in the intervention and 120 in the comparison group.

Inclusion criteria Adults 18 years and older with confirmed T2D (as diagnosed by physicians and based on the history of medicines they have been taking) Exclusion criteria Patients with diabetes type 1, gestational diabetes, pregnant women and people with severe cognitive impairment or terminally ill people Intervention Training handbook For a phased and an intensified DSME, an Ethiopian context patient friendly handbook with illustrative pictures has been prepared. To help illiterate/less-literate patients the DSME materials are mainly supported by illustrative pictures with short text explanations. The content includes: basics of diabetes, healthy eating, healthy exercise, medication management, prevention of acute and long-term complications, foot care and psychosocial issues in diabetes.

For contextualization appropriate expertise like physicians, nurses, pharmacists, linguistics and others were consulted. All the DSME materials were translated in to Amharic and Afan Oromoo languages.

Provider The DSME sessions have been given by the PhD student and a clinical nurse who has experience of working with diabetes patients and is fluent in Afan Oromo and Amharic. The nurse was trained for a total of 16 hours before starting the education session.

Duration Participants enrolled in the intervention group sessions of have got DSME every month on their date of appointment for six consecutive months for a total of approximately 9 hours. For convenience all the sessions will be held on the date of their routine follow-up before seen by doctors.

Approach Each of the six sessions was interlinked with take home activities and experience sharing in the subsequent session. The first five sessions was framed with specific areas of discussion, whereas the sixth (last) session will be revision through sharing their experiences over the last five months. After the six sessions were addressed over six months, the intervention group was followed for the next three consecutive months with brief sessions of discussion. The comparison group continued getting the usual care.

The approach of the DSME sessions focused on experience sharing where patients share their experiences of diabetes management, daily life, life-style modification, complication risk reduction, etc. which is supported by education sessions.

Data Collection Tool and Technique At base line data was collected from both intervention and comparison groups. Then, three months after completion of DSME end-line survey will be conducted.

For base line data collection interview of patients, record review, anthropometric measurements, and laboratory tests were used. Before data collection those doing interview, taking anthropometric measurements, and taking blood samples were trained for one day.

Data related to socio-demographic characteristics, food security, diabetes self-care practice, medication adherence, health care utilization, BP, weight, height, WC, BGL, HbA1c, HRQoL, self-efficacy, depression, stress and diabetes knowledge were collected at baseline and follow-up surveys. In addition, at the end of the intervention patients' feeling about the overall DSME sessions will be elicited. Key points from the group discussions have been recorded by the PhD student.

This project is being undertaken in a resource limited facility where laboratory facility is limited, bureaucracy or uncooperativeness of administrative bodies and different members of health care team may happen to use existing laboratory services for the end-line survey.

Pilot All of questionnaires/tools was translated to Amharic and Afan Oromo and then back translated to English. Before the actual intervention and baseline survey a pilot study was conducted on a 5% of the study population to customize the questionnaires to the Ethiopian context. Based on findings from the pilot, appropriate amendments were made.

Analysis Descriptive statistics will be used as required. Chi-square tests will be employed to compare the intervention and comparison groups, in terms of the components of outcomes. Logistic regression will be employed to determine factors affecting the implementation of DSME. Intension to treat analysis will be used for the analysis of the outcome variables.

Regarding qualitative data from each group discussions, key data will be summarized, and analysis of comments or quotes of participants will be labeled for analysis by theme.

Research Ethics Before the commencement of the study, ethical approval letters were secured from REK (Norwegian Regional Committee for Medical and Health Research Ethics) and Jimma University Ethical Review Board. Moreover, at the level of recruitment a written consent was secured from each study participant.

Since the aim of the study is to determine the effect of DSME, the comparison group didn't get education. Nevertheless, like the intervention group their blood glucose have been tested on every visit. Moreover, during base line survey any question that the comparison group members asked have been explained, which will be similar on the end-line survey too.

Blood samples and data that are registered about the patient only be used in accordance with the purpose of the study. On base line blood sample collected for BGL and HbA1c was discarded immediately after the analysis procedure. Similarly on the end-line survey blood samples will be discarded immediately after the test is done. All the data and samples are being processed without name, ID number or other directly recognizable type of personal information. A code number links the specific patient to his/her data and samples through a list of names. Only authorized project personnel have access to the list of names and be able to identify the patient. All data is stored in Services for Sensitive Data (TSD) server of University of Oslo. It will not be possible to identify individual patient in published or presented results from the study. All data will be discarded five years after the end of the project.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older with confirmed T2DM (as diagnosed by physicians and based on the history of medicines they have been taking) were recruited. People with T2DM and other co-morbid diseases like cardiovascular diseases were included.

Exclusion Criteria:

* Patients with diabetes type 1, gestational diabetes, pregnant women and people with severe cognitive impairment or terminally ill people were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Proportion of T2D patients with controlled BGL as measured by a change in HbA1c | HbA1c was measured on baseline, which was done 5 months before the commencement of the intervention. A change in HbA1c will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  The glycemic control is measured by the level of HbA1c where HbA1c>=7% indicates poorly controlled diabetes and <7% well controlled roughly over the last three months

SECONDARY OUTCOMES:
Proportion of T2D patients with a recommended level of diabetes self-care behavior as measured by summary of diabetes self-care activities (SDSCA) questionnaire | Proportion of T2D patients with the recommended level of diabetes self-care behavior was measured on baseline. Behavioral change will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  Diabetes self-care activities related to self-care practices that include healthy eating, physical exercise, blood sugar monitoring, medication adherence, foot care and smoking

OTHER OUTCOMES:
change in health related quality of life (HRQoL) | HRQoL over the last 24 hours was measured on baseline. A change in HRQoL over the last 24 hours will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  Intended to measure the effect of the educational session on the overall health status of patients as measured by four items howRu quality assessment tool over the last 24 hours
Level of diabetes management knowledge as measured by true/false form of simplified diabetes knowledge questionnaire (SDKS). | Diabetes management knowledge was measured on baseline and a change in diabetes management knowledge will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  Diabetes is intended to measure the effect of the educational session on their knowledge of diabetes management as measured by SDKS which is a simplified form of diabetes knowledge assessment tool recommended for less literate study participants.
Level of confidence in performing diabetes self-care behaviors as measured by Diabetes Self-Efficacy Scale developed by Standford Patient Education Research Center | Level of confidence in performing diabetes self-care behaviors was measured on baseline. A change in level of confidence will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  Self-efficacy is intended to measure how effective an intensified DSME session is on patients confidence in performing self-care activities like confidence in food selection, food preparation, diabetes control, etc
Change in the level of perceived stress as measured by global measure of perceived stress | Level of perceived stress was measured on baseline and a change in level of perceived stress will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  It is intended to measure how effective an intensified DSME session is in reducing level of stress among diabetes patients, which is measured by global measure of perceived stress tool which has got 14 items
Change in the level of depressive symptoms as measured by patient health questionnaire depression scale (PHQ-9) | Level of depressive symptoms was measured on baseline and a change in level of depressive symptoms will be measured 9 months after the commencement of the intervention or 14 months after commencement of the intervention.
  It is intended to measure how effective an intensified DSME session is in reducing depressive symptoms among diabetes patients which is measured by the 9-items PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Fikadu B Hailu, PhD Fellow, Principal Investigator — Jimma University; Anne Moen, PhD, Study Chair — University of Oslo; Per Hjortdahl, PhD, Study Director — University of Oslo

IPD SHARING:
Plan to Share IPD: Yes
For researchers interested in the area of DSME individual participant data (IPD) will be available to them with official request. Before sharing all members of research, team will be consulted and any data indicating participants' identification will be exempted. In case a part of raw data is requested as a secondary data for further analysis and publication it will be made with the active involvement of all research team members.

REFERENCES:
- [Background] Mendis S, Davis S, Norrving B. Organizational update: the world health organization global status report on noncommunicable diseases 2014; one more landmark step in the combat against stroke and vascular disease. Stroke. 2015 May;46(5):e121-2. doi: 10.1161/STROKEAHA.115.008097. Epub 2015 Apr 14. No abstract available. PMID 25873596
- [Background] Barr VJ, Robinson S, Marin-Link B, Underhill L, Dotts A, Ravensdale D, Salivaras S. The expanded Chronic Care Model: an integration of concepts and strategies from population health promotion and the Chronic Care Model. Hosp Q. 2003;7(1):73-82. doi: 10.12927/hcq.2003.16763. PMID 14674182
- [Background] Idemyor V. Diabetes in sub-Saharan Africa: health care perspectives, challenges, and the economic burden of disease. J Natl Med Assoc. 2010 Jul;102(7):650-3. doi: 10.1016/s0027-9684(15)30643-x. PMID 20690330
- [Background] Peer N, Kengne AP, Motala AA, Mbanya JC. Diabetes in the Africa Region: an update. Diabetes Res Clin Pract. 2014 Feb;103(2):197-205. doi: 10.1016/j.diabres.2013.11.006. Epub 2013 Dec 1. PMID 24315460
- [Background] Beran D. The Diabetes Foundation Report on implementing national diabetes programmes in sub-Saharan Africa, 2006. International Insulin Foundation: London.
- [Background] Beran D, Yudkin JS. Diabetes care in sub-Saharan Africa. Lancet. 2006 Nov 11;368(9548):1689-95. doi: 10.1016/S0140-6736(06)69704-3. PMID 17098088
- [Background] Snoek Fj, Visser A. Improving quality of life in diabetes: how effective is education? Patient Educ Couns. 2003 Sep;51(1):1-3. doi: 10.1016/s0738-3991(03)00204-0. No abstract available. PMID 12915274
- [Background] Tuei VC, Maiyoh GK, Ha CE. Type 2 diabetes mellitus and obesity in sub-Saharan Africa. Diabetes Metab Res Rev. 2010 Sep;26(6):433-45. doi: 10.1002/dmrr.1106. PMID 20641142
- [Background] Fisher EB, Boothroyd RI, Coufal MM, Baumann LC, Mbanya JC, Rotheram-Borus MJ, Sanguanprasit B, Tanasugarn C. Peer support for self-management of diabetes improved outcomes in international settings. Health Aff (Millwood). 2012 Jan;31(1):130-9. doi: 10.1377/hlthaff.2011.0914. PMID 22232103
- [Background] MakkiAwouda FO, Elmukashfi TA, Hag Al-Tom SA. Effects of health education of diabetic patient's knowledge at Diabetic Health Centers, Khartoum State, Sudan: 2007-2010. Glob J Health Sci. 2014 Feb 14;6(2):221-6. doi: 10.5539/gjhs.v6n2p221. PMID 24576384
- [Background] Mash RJ, Rhode H, Zwarenstein M, Rollnick S, Lombard C, Steyn K, Levitt N. Effectiveness of a group diabetes education programme in under-served communities in South Africa: a pragmatic cluster randomized controlled trial. Diabet Med. 2014 Aug;31(8):987-93. doi: 10.1111/dme.12475. Epub 2014 May 20. PMID 24766179
- [Derived] Hailu FB, Moen A, Hjortdahl P. Diabetes Self-Management Education (DSME) - Effect on Knowledge, Self-Care Behavior, and Self-Efficacy Among Type 2 Diabetes Patients in Ethiopia: A Controlled Clinical Trial. Diabetes Metab Syndr Obes. 2019 Nov 29;12:2489-2499. doi: 10.2147/DMSO.S223123. eCollection 2019. PMID 31819574
- [Derived] Hailu FB, Hjortdahl P, Moen A. Nurse-Led Diabetes Self-Management Education Improves Clinical Parameters in Ethiopia. Front Public Health. 2018 Oct 23;6:302. doi: 10.3389/fpubh.2018.00302. eCollection 2018. PMID 30406070
- See also: Global status report on noncommunicable diseases 2010 — http://apps.who.int/iris/bitstream/10665/44579/1/9789240686458_eng.pdf
- See also: Type 2 diabetes mellitus and obesity in sub-Saharan Africa — http://onlinelibrary.wiley.com/doi/10.1002/dmrr.1106/pdf
- See also: Effects of Health Education of Diabetic Patient's Knowledge at Diabetic Health Centers, Khartoum State, Sudan: 2007-2010 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4825225/
- See also: Educational and Psychological Issues Effectiveness of a group diabetes education programme in under-served communities in South Africa: a pragmatic cluster randomized controlled trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4232864/pdf/dme0031-0987.pdf
- See also: Determinants of glycemic control among insulin treated diabetic patients in Southwest Ethiopia: hospital based cross sectional study. — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0061759